CLINICAL TRIAL: NCT01597336
Title: Treatment of Abdominal Abscesses With or Without Fibrinolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11120126
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Abdominal Abscess; Tissue Plasminogen Activator
Keywords: abscess; tPA
MeSH Terms: conditions — Abdominal Abscess; Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline only flush of abscess (Active Comparator): Saline alone used to flush abscess
  Interventions: Procedure: Saline flush of abscess
- Saline plus tPA flush of abscess (Experimental): Saline plus tPA used for abscess flush
  Interventions: Procedure: Tissue plasminogen activator abscess flush

INTERVENTIONS:
Procedure: Tissue plasminogen activator abscess flush — Thirteen ml of 10% tPA in saline at time of drain and twice daily thereafter.
  Other Names: fibrinolytic abscess flush
  Arms: Saline plus tPA flush of abscess
Procedure: Saline flush of abscess — Thirteen ml of saline is used to flush abscess at time of drain placement and twice daily thereafter.
  Other Names: Standard saline flush of abscess
  Arms: Saline only flush of abscess

SUMMARY:
The objective of this study is to evaluate the utility of fibrinolysis when draining an abdominal abscess as defined by length of stay after drainage.

DETAILED DESCRIPTION:
The hypothesis is that fibrinolysis of a abscess will shorten hospital stay compared to drainage alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients under age 18 found to have an abscess in their abdomen related to perforated appendicitis that requires a drain either prior to or after appendectomy.

Exclusion Criteria:

* Patients with known immune deficiency per medical record review
* Patients with another condition affecting surgical decision making or recovery
* Patients with drain unable to be placed

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 1-2 weeks
  Length of time required for meeting discharge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States